CLINICAL TRIAL: NCT00077584
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Study to Assess the Effect of Bosentan on Healing and Prevention of Ischemic Digital Ulcers in Patients With Systemic Sclerosis
Brief Title: Efficacy and Safety of Oral Bosentan on Healing/Prevention of Digital (Finger) Ulcers in Patients With Scleroderma
Acronym: RAPIDS-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-052-331; NCT02800993 (obsolete NCT alias)
Record Dates: First submitted 2004-02-10; First posted 2004-02-11 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Digital Ulcers; Systemic Sclerosis
Keywords: Scleroderma; Finger Ulcers; Digital Ulcers; Systemic Sclerosis
MeSH Terms: conditions — digital ulcers; Scleroderma, Systemic; Scleroderma, Diffuse | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Bosentan (Experimental): The patients received bosentan 62.5 mg twice daily (b.i.d.) for 4 weeks and then 125 mg b.i.d. for 20 weeks
  Interventions: Drug: Bosentan 62.5 mg; Drug: Bosentan 125 mg
- Placebo (Placebo Comparator): The patients received the matching placebo for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bosentan 62.5 mg — Oral tablets containing 62.5 mg of bosentan
  Other Names: Ro 47-0203
  Arms: Bosentan
Drug: Bosentan 125 mg — Oral tablets containing 125 mg of bosentan
  Other Names: Ro 47-0203
  Arms: Bosentan
Drug: Placebo — Oral tablets matching bosentan 62.5-mg tablets and bosentan 125-mg tablets
  Arms: Placebo

SUMMARY:
In an earlier clinical trial, RAPIDS-1, conducted in scleroderma patients with or without digital ulcers at baseline, bosentan significantly reduced the number of new digital ulcers versus placebo. The purpose of the present trial (RAPIDS-2) is to evaluate the prevention and healing effects of bosentan versus placebo on digital ulcers over a 24-week treatment period.

ELIGIBILITY:
Main Inclusion Criteria:

* Systemic Sclerosis (SSc), diffuse or limited.
* SSc patients with at least one digital ulcer at baseline qualifying as a cardinal ulcer.

Main Exclusion Criteria:

* Digital ulcers due to conditions other than SSc.
* Severe pulmonary arterial hypertension (PAH) (Who class III and IV).
* Malabsorption or any severe organ failure (e.g., lung, kidney, liver) or any life-threatening condition.
* Treatment with parenteral prostanoids (prostaglandin E, epoprostenol, or prostacyclin analogs) during the past 3 months prior to randomization.
* Treatment with inhaled or oral prostanoids one month prior to randomization.
* Previous treatment with bosentan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2003-10; Primary Completion 2005-03 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Time to complete healing of the cardinal ulcer (CU) up to Week 24 in patients with CU healing maintained for 12 weeks | 24 weeks
Total number of new digital ulcers per patient up to Week 24 | 24 weeks

SECONDARY OUTCOMES:
Change from baseline to Week 24 in hand pain | Baseline and Week 24
  Pain assessed on visual analog scales
Change from baseline to Week 24 in hand disability | Baseline and Week 24
  Hand disability indexed assessed using the Health Assessment Questionaire (HAQ)
Proportion of subjects with treatment-emergent adverse events | up to 32 weeks (8 week post-treatment follow-up)
Proportion of subjects with liver function abnormalities | Every 4 weeks up to Week 24
  Increase in aminotransferases

CONTACTS AND LOCATIONS:
Overall Officials: James Seibold, MD, Principal Investigator — Robert Wood Johnson Medical School, New Brunswick, NJ, USA

REFERENCES:
- [Result] Matucci-Cerinic M, Denton CP, Furst DE, Mayes MD, Hsu VM, Carpentier P, Wigley FM, Black CM, Fessler BJ, Merkel PA, Pope JE, Sweiss NJ, Doyle MK, Hellmich B, Medsger TA Jr, Morganti A, Kramer F, Korn JH, Seibold JR. Bosentan treatment of digital ulcers related to systemic sclerosis: results from the RAPIDS-2 randomised, double-blind, placebo-controlled trial. Ann Rheum Dis. 2011 Jan;70(1):32-8. doi: 10.1136/ard.2010.130658. Epub 2010 Aug 30. PMID 20805294
- [Derived] Liu C, Chen J, Gao Y, Deng B, Liu K. Endothelin receptor antagonists for pulmonary arterial hypertension. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD004434. doi: 10.1002/14651858.CD004434.pub6. PMID 33765691